CLINICAL TRIAL: NCT02626260
Title: A Pilot Evaluation of Adhesives and How They Are Impacted by Output
Brief Title: A Pilot Evaluation of Adhesives and How They Are Impacted by Output (Round 1b)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_01b
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2017-08

CONDITIONS: Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1b (Experimental): The subject test one adhesive strip on the peristomal area
  Interventions: Other: adhesive strip

INTERVENTIONS:
Other: adhesive strip — Adhesive strip with a standard adhesive base

SUMMARY:
The study investigates the impact real output has on the adhesion of adhesives.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Remaining adhesive area of adhesive | 30 hours
  The remaining adherent area of the adhesive is assessed by subtracting the area of output and swelling from the total adhesive area

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark